CLINICAL TRIAL: NCT00901056
Title: Feasibility Study to Investigate the Effect of Low Intensity Shockwaves on Patients With Erectile Dysfunction Resulted From Vascular Origin
Brief Title: Extracorporeal Shock Wave Therapy for the Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medispec (Industry)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Prof. Yoram Vardi, Rambam Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ED-ESWT
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-11

CONDITIONS: Erectile Dysfunction
Keywords: ED; Erectile Dysfunction; Erectile dysfunction treated with PDE-5 inhibitors
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated Group (Active Comparator): This group will receive actual shockwave treatment
  Interventions: Device: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy — Energy Density - 0.02 - 0.15 mJ/mm2
  Other Names: Vascuspec

SUMMARY:
Low intensity shockwaves have been proven in animal studies to induce local growth of new blood vessels from existing ones.

The hypothesis of this study is that shockwave therapy could improve the symptoms of patients with erectile dysfunction resulted from a vascular origin and respond to PDE-5 inhibitors.

DETAILED DESCRIPTION:
Low intensity shockwaves (1/10 the ones used in Lithotripsy) are delivered to the penile tissue. Shockwaves are created by a special generator and are focused using a specially designed shockwave applicator apparatus. The shockwaves are delivered trough the applicator covering the corpora cavernosa of the penis.

ELIGIBILITY:
Inclusion Criteria:

* ED of more than 6 months
* At least 50% unsuccessful to attempt sexual intercourse for 4 times at 4 different days
* Positive response to PDE-5 inhibitors
* IIEF-5 domain score of 12-20 denoting mild to severe ED
* Non-Neurological pathology
* Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* NPT - normal/flat
* Prior prostatectomy surgery
* Any cause of ED other than vascular related
* Any unstable medical, psychiatric, spinal cord injury, penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Cardiovascular conditions that prevent sexual activity
* History of heart attack, stroke or life-threatening arrhythmia within the prior 6 months.
* Cancer within the past 5 years.
* Anti-androgens, oral or injectable androgens
* Use of any treatment for ED within 7 days of screening including oral medications, vacuum devices, constrictive devices, injections or urethral suppositories

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
IIEF score | 3 months

SECONDARY OUTCOMES:
Rigid Score (RS) | 3 months
Quality of Erection Questionnaire (QEQ) | 3 months
Self-Esteem And Relationship Questionnaire (SEAR) | 3 months
Erectile Dysfunction Inventory of Treatment Satisfaction (EDIT) | 3 months
Side Effects | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Vardi, Professor, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel